CLINICAL TRIAL: NCT05648656
Title: Efficacy of TXA Nebulization for the Treatment of Hemoptysis: A Randomized Controlled Clinical Trial
Brief Title: TXA Nebulization for the Treatment of Hemoptysis
Acronym: TXA-NEB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Deba Prasad Dhibar, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INT/IEC/2021/SPL-1634
Record Dates: First submitted 2022-12-02; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Hemoptysis
MeSH Terms: conditions — Hemoptysis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TXA (Active Comparator): Nebulization with TXA 500mg/ 5mL 8 hourly for 2 days.
  Interventions: Drug: TXA Nebulization
- Control (Placebo Comparator): Nebulization with 0.9%normal saline 5mL 8 hourly for 2 days
  Interventions: Other: 0.9% NS Nebulization

INTERVENTIONS:
Drug: TXA Nebulization — Nebulization with TXA 500mg/ 5mL 8 hourly for 2 days plus standard care of therapy
  Arms: TXA
Other: 0.9% NS Nebulization — Nebulization with 0.9% normal saline (NS) 5mL 8 hourly for 2 days plus standard care of therapy
  Arms: Control

SUMMARY:
Hemoptysis is a common presentation in medical emergency. Prompt medical therapy, bronchoscopic and endovascular procedures remains the cornerstone of management for both diagnostic as well as therapeutic purpose in hemoptysis. Priority is given for medical management to achieve hemostasis and prevent aspiration as well as treatment of underlying etiology, before undertaking any definitive bronchoscopic or endovascular intervention. While majority of the patients are managed successfully by prompt medical therapy, only the refractory cases and life-threatening hemoptysis need more definitive procedures like DSA guided bronchial artery embolization and bronchoscopic procedures like endobronchial biocompatible glue, endobronchial embolization using silicone spigots, endobronchial stents, laser photocoagulation. Tranexamic acid is an anti-fibrinolytic agent which prevent breakdown of fibrin clots, thus helping in clot stabilization and controlling bleeding. As a medical therapy Tranexamic Acid is used for bleeding control in hemoptysis as well as other surgical or traumatic bleeding. Previously conducted institutional study comparing IV infusion of TXA to placebo in patients with sub massive hemoptysis showed results favoring TXA over placebo in terms of decreasing frequency & quantity of hemoptysis, duration of hospital stay and need for DSA/ broncoscopic/ surgical intervention and blood transfusion (1). While the oral and IV routes have been most commonly studied, use of novel approaches like aerosolized TXA and endobronchial instillation of TXA during bronchoscopy have showed positive results in achieving hemostasis in hemoptysis (2). A recently conducted RCT, to assess the effectiveness of TXA nebulization in sub-massive hemoptysis concluded that nebulized TXA is effective in reducing the frequency and quantity of hemoptysis. Nebulized TXA was also found to be safe as no severe ADR was noted during its use as per previous RCT as well as multiple case reports.

However, because of limited number of research with small sample size and barring some case reports evidence for the use of nebulized TXA is limited in hemoptysis. In hemoptysis nebulized form of TXA is supposed to reach local site of bleeding (lung/ airway) promptly at a higher concentration leading to rapid control of hemoptysis. So, this study has been planned to evaluate further this novel approach of TXA nebulization for the management of hemoptysis. Similarly, data regarding adverse drug reaction related to TXA nebulization is also limited. This study will produce additional information regarding efficacy, safety and ADR related to TXA nebulization.

ELIGIBILITY:
Inclusion Criteria:

* All cases of active hemoptysis
* irrespective of gender
* age≥ 18 years

Exclusion Criteria:

* Massive hemoptysis
* Pregnancy
* Drug allergy to TXA4
* Renal failure
* Receiving Oral Contraceptive Pills.
* Already on blood thinner
* Not willing for consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of hemoptysis | 48 hours
  Number of episode of hemoptysis per day will be compared at baseline and day 2 (48 hours)
Quantity of hemoptysis | 48 hours
  Through collection of expectorated blood, quantityofhemoptysis per day will be compared at baseline and day2 (48hours) .
Visual analogue scale (VAS) | 48 hours
  Visual subjective assessment by the patient will be used to compare the amount of hemoptysis at baseline and day 2 (48 hours). VAS will be presented to the patients as a 100 mm line anchored by description with 'no-hemoptysis' at one end and 'worst imaginable hemoptysis' on the other end. Patients will be asked to mark a point on the 100 mm line to indicate the severity.
  A millimeter scale will be used to measure the score and this will provide 0-100 levels of hemoptysis and the score increases with increasing severity.

SECONDARY OUTCOMES:
Adverse drug events | 48 hours
  Frequency/number of adverse drug events will be compared between the groups.
Resolution of hemoptysis | 48 Hours
  Resolution of hemoptysis is defined as no episode of hemoptysis containing fresh blood sustained for at least 48 hours following cessation of hemoptysis. The rate of resolution of hemoptysis will be compared between the groups.
Need for intervention | 48 Hours
  The overall the rate of the need for therapeutic interventional procedures (BAE, bronchoscopic procedures), to achieve hemostasis, will be compared between the study and control group.
Need for blood transfusion | 48 Hours
  The percentage of patients requiring blood transfusion as well as the mean number of PRBCs transfused will be compared between the groups.
Duration of hospital stay | 4 weeks
  The total duration of hospital stay (from the day of admission to the day of discharge or death) will be compared between both the groups.
Mortality | 4 weeks
  All patients will be followed up at day 28, physically or telephonically to assess the mortality as well as their well-being. The rate of mortality will be compared between the groups.
Recurrence of hemoptysis | 4 weeks
  Recurrence will be defined as fresh episode of hemoptysis after resolution during 28 days follow-up. The rate of recurrence of hemoptysis will be compared between the groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agrawal A, Dhibar DP, Prakash A, Sreedhara BC, Muthu V, Pannu AK. Efficacy and safety of tranexamic acid nebulization to control bleeding of hemoptysis: The TXA-NEB randomized controlled clinical trial. Indian J Pharmacol. 2025 Nov 1;57(6):392-400. doi: 10.4103/ijp.ijp_824_25. Epub 2025 Oct 12. PMID 41221568